CLINICAL TRIAL: NCT00454441
Title: Sleep Quality in CHIMES (MF101)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bionovo (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: MF101 Ancillary Study
Record Dates: First submitted 2007-03-28; First posted 2007-03-30 (Estimated); Last update posted 2007-03-30 (Estimated); Status verified 2007-03

CONDITIONS: Sleep Quality; Menopausal Symptoms
Keywords: Sleep Quality; Menopausal Symptoms; Actigraph; Bionovo; MF101
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

INTERVENTIONS:
Drug: MF101

SUMMARY:
Menopausal women often complain of difficulty sleeping and the transition from pre- to postmenopausal status is associated with an incresase in self-reported sleep disturbance. Hot flashes have been associated with self-reported measures of sleep disturbance and changes in sleep pattern as measured by plysomnography, including an increase in stage 4 and a latency or shortened time in rapid-eye movement sleep. Although there are some data on the effect of hormone replacement therapy on self-reported sleep measures in symptomatic postmenopausal women, there are no data on the effect of herbal extracts on subjective or objective measures of sleep quality in this population group. Actigraphy, the use of a device to record movement generally placed on the wrist, has been used over 20 years to provide objective data concerning sleep/wake patterns. The advantage of actigraphy over traditional polysomnography is that actigraphy can conveniently record continuously for 24-hours a day for longer periods of time.

DETAILED DESCRIPTION:
Specific Aims:

1. To determine the effect of MF101 (a combination of Chinese herbs) compared to placebo on change in sleep quality utilizing baseline and follow-up actigraphy obtained from a subset of approximately 90 women enrolled in the randomized, double-blind, placebo-controlled Chinese Herbs for Menopausal Symptoms (CHIMES) trial.
2. TO identify the correlates of sleep quality as assessed by actigraphy in women with frequent hot flashes. We will evaluate demographic, lifestyle, anthropometric, medical and gynecologic history and hormonal factors that may relate to the actigraphic measures of sleep quality, including self-reported measures of sleep.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 40 to 60.
* Currently receiving medical care from a health care provider.
* Self-report 5 hot flashes per day or 35 hot flashes per week.
* Postmenopausal as defined by 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels > 30mlU/ml or 6 weeks post-surgical bilateral oophorectomy with or without hysterectomy or hysterectomy with FSH levels > 30 mlU/ml.
* Agree not to start new herbal or dietary supplements and not to change the dose of any currently used herbal or dietary supplements for the duration of the trial.
* Successful completion of a Hot Flash Diary, a Daily Study Medication Diary and a Bleeding Diary, tolerates placebo, and 80% compliant at run-in.
* Must have had a mammogram within the last 9 months.
* Have access to a phone.
* Provide informed consent.

Exclusion Criteria:

* Inability to sign an informed consent or fill out questionnaires.
* History of breast, uterine or ovarian cancer or melanoma.
* Abnormal mammogram or breast examination within the last 9 months suggestive of cancer.
* Abnormal Pap smear or pelvic examination within the last 9 months suggestive of cancer.
* Double-wall endometrial thickness that exceeds 5 mm measured on transvaginal ultrasound.
* Unexplained abnormal uterine bleeding within six months of enrollment.
* Pregnancy or lactating.
* Clinical evidence of active ischemic cardiovascular disease or a history of cardiovascular disease.
* History of deep vein thrombosis or pulmonary embolism requiring anticoagulation.
* Active liver or gallbladder disease.
* Use of medications, herbal or dietary supplements known to possibly be effective for the treatment of hot flashes within three months of enrollment for oral or transdermal drugs, or within 6 months of enrollment for implanted or injected drugs.
* Use of raloxifene or tamoxifen within three months of enrollment.
* Use of another investigational agent within 3 months of enrollment.
* History of multiple or severe food or medicine allergies.
* Any medical or psychiatric condition that, in the investigator's opinion, would preclude the participant from adhering to the protocol or completing the trial, including severe illness, plans to move, substance abuse, significant problems, or dementia.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180
Dates: Start 2006-02; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Actigraph watch (SleepWatch-O, Ambulatory Monitoring, Inc., Ardsley, NY)

CONTACTS AND LOCATIONS:
Overall Officials: Kristine Ensrud, MD, MPH, Principal Investigator — University of Minnesota Twin Cities Campus
Locations (2):
- United States (2):
  - University of California, San Francisco, San Francisco, California
  - University of Minnesota Twin Cities Campus, Minneapolis, Minnesota